CLINICAL TRIAL: NCT05699525
Title: Efficacy of Personalized Mobile Cognitive Behavioral Therapy Targeting Anxiety and Depression
Brief Title: Personalized Mobile Cognitive Behavioral Therapy Application
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Children's Health Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-09023953
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders and Symptoms; Depression; Bipolar Disorder; Symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression; Bipolar Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized (Experimental): Participants receive the personalized Maya app intervention for 6 weeks
  Interventions: Behavioral: Personalized MAYA Mobile App
- General Non-Personalized (Active Comparator): Participants receive the general MAYA app intervention for 6 weeks
  Interventions: Behavioral: General MAYA Mobile App

INTERVENTIONS:
Behavioral: Personalized MAYA Mobile App — All new material in the personalized condition will be introduced within the first four weeks and will contain modules targeting participant's personal symptom profiles. The remaining two weeks in the personalized condition will consist of practicing previously learned skills.
  Arms: Personalized
Behavioral: General MAYA Mobile App — New material will be introduced to participants over all the six weeks of the intervention and will include all application modules.
  Arms: General Non-Personalized

SUMMARY:
This study aims to compare the effectiveness of a standard mobile iPhone cognitive behavioral therapy program to a personalized mobile iPhone cognitive behavioral therapy program that introduces new skills over a shorter period of time. Participants will use the Maya app for two days per week, at least 20 minutes per day, for six weeks. Assessments will include a weekly check in with a member of the research team, questionnaires, and optional magnetic resonance imaging (MRI) and electroencephalographic (EEG) recordings at the beginning and end of the 6-week intervention. The investigators think that that the less burdensome personalized program will be just as effective at improving symptoms of anxiety and depression as the general program.

DETAILED DESCRIPTION:
Growing evidence suggests a need for anxiety and mood interventions that can be disseminated easily to adolescents and young adults. The goal of this study is to optimize a mobile application that teaches well-established, research-supported psychotherapeutic techniques to adolescents and young adults who are experiencing symptoms of anxiety, depression, and/or bipolar disorder. The study aims to compare the efficacy of a personalized mobile cognitive behavioral therapy program to a more general mobile cognitive behavioral therapy program.

Study participants will randomly receive one of two versions of Maya, a mobile cognitive behavior therapy (CBT) app for adolescents and young adults: either a standard version that includes a variety of skills typically used in CBT, or a personalized version with skills matched to the participant's symptom profile. In contrast to the general condition, which may introduce new material over all six weeks of the intervention, all new material in the personalized condition will be introduced within the first four weeks. The remaining two weeks in the personalized condition will consist of practicing previously learned skills. Participants will use the Maya app for two days per week, at least 20 minutes per day for six weeks and will complete assessments at baseline, week 4, week 6 (end of intervention), and a follow-up assessment at week 12. Participants may also choose to complete an optional magnetic resonance imaging (MRI) and/or electroencephalographic (EEG) recording at the baseline and end of intervention (week 6).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years.
* Primary diagnosis of an anxiety, depressive, or bipolar disorder as determined by a score of 4 or greater on the Clinical Severity Rating of the Anxiety Disorders Interview Schedule (ADIS).
* If an individual is diagnosed with bipolar disorder, they must be currently euthymic or experiencing a depressive episode.
* Access to an Apple iPhone

Exclusion Criteria:

* History of neurologic disorder that may affect the neural systems of interest or participant's ability to participate
* Lifetime diagnosis of a psychotic disorder.
* Current hypomanic or manic episode.
* Currently in cognitive behavior therapy.
* Change in dose of a psychiatric medication in the past 12 weeks.
* Initiation of psychotherapy in the past 12 weeks.
* Intent or plan to attempt suicide.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms from pre-intervention to post-intervention as measured by the HAM-A. | Baseline to endpoint [Week 6]
  The primary symptom measure for anxiety will be the Hamilton Rating Scale for Anxiety (HAM-A). The HAM-A is a 14-item questionnaire measure of the severity of anxiety symptoms. The items measure both psychic anxiety and somatic anxiety. The scores range from 0 to 56, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no anxiety symptoms.
Change in depressive symptoms from pre-intervention to post-intervention as measured by HAM-D. | Baseline to endpoint [Week 6]
  The primary symptom measure for depression will be the Hamilton Rating Scale for Depression (HAM-D). The HAM-D is a 24-item questionnaire measuring the severity of depression symptoms. The scale ranges from 0 to 76, where higher scores indicate higher severity of depressive symptoms.
Change in anxiety symptoms from pre-intervention to post-intervention as measured by the anxiety subscale of the DASS. | Baseline to endpoint [Week 6]
  Anxiety will be measured by the anxiety subscale of the Depression Anxiety Stress Scale (DASS). The anxiety subscale measures of the severity of anxiety symptoms. The scores range from 0 to 42, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no anxiety symptoms.
Change in depressive symptoms from pre-intervention to post-intervention as measured by the depression subscale of the DASS. | Baseline to endpoint [Week 6]
  Depression will be measured by the depression subscale of the Depression Anxiety Stress Scale (DASS). The subscale measures of the severity of depressive symptoms. The scores range from 0 to 42, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no symptoms.

SECONDARY OUTCOMES:
Change in anxiety measure scores pre-intervention to post-active learning phase as measured by HAM-A | Baseline to end of active learning phase [week 4]
  Anxiety will be measured using the Hamilton Rating Scale for Anxiety (HAM-A). The HAM-A is a 14-item questionnaire measure of the severity of anxiety symptoms. The items measure both psychic anxiety and somatic anxiety. The scores range from 0 to 56, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no anxiety symptoms.
Change in anxiety measure scores pre-intervention to post-active learning phase as measured by the anxiety subscale of the DASS. | Baseline to end of active learning phase [week 4]
  Anxiety will be measured by the anxiety subscale of the Depression Anxiety Stress Scale (DASS). The anxiety subscale measures of the severity of anxiety symptoms. The scores range from 0 to 42, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no anxiety symptoms.
Change in depression measure scores pre-intervention to post-active learning phase as measured by HAM-D. | Baseline to end of active learning phase [week 4]
  Depression will be scored using the Hamilton Rating Scale for Depression (HAM-D). The HAM-D is a 24-item questionnaire measuring the severity of depression symptoms. The scale ranges from 0 to 76, where higher scores indicate higher severity of depressive symptoms.
Change in depression measure scores pre-intervention to post-active learning phase as measured by the depression subscale of the DASS. | Baseline to end of active learning phase [week 4]
  Depression will be measured by the depression subscale of the Depression Anxiety Stress Scale (DASS). The subscale measures of the severity of depressive symptoms. The scores range from 0 to 42, where higher scores indicate a greater severity of symptoms and lower scores indicate mild to no symptoms.
Change in social anxiety from pre-intervention to post-intervention as measured by LSAS. | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Social anxiety will be measured using the Liebowitz Social Anxiety Scale (LSAS). The items measure social anxiety and extent of avoidance. Scores range from 0 to 144 where higher scores indicate higher levels of social anxiety.
Change in anxiety sensitivity from pre-intervention to post-intervention as measured by ASI. | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Anxiety sensitivity will be measured using the Anxiety Sensitivity Index (ASI). The items measure distress intolerance and fear of anxiety related sensations. Scores range from 0 to 72 where higher scores indicate higher levels of anxiety sensitivity.
Change in avoidance from pre-intervention to post-intervention as measured by MEAQ. | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Experiential avoidance will be measured using the Multidimensional Experiential Avoidance Questionnaire (MEAQ). The 62-item scale measures avoidance of negative internal experiences. Scores range from 62 to 372 where higher scores indicate higher levels of anxiety sensitivity.
Change in anhedonia from pre-intervention to post-intervention as measured by TEPS. | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Anhedonia will be measured using the Temporal Experience of Pleasure Scale (TEPS). The items measure anticipatory and consummatory experiences of pleasure. Scores range from 18 to 108 where higher scores indicate stronger feelings of anticipating and experiencing pleasure.
Change in Negative affect from pre-intervention to post-intervention as measured by PANAS | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Negative affect will be measured using the negative affect subscale of the Positive and Negative Affect Schedule (PANAS). Scores on the 10-item subscale range from 10 to 50, where higher scores indicate higher levels of negative affect.
Bipolar symptoms from pre-intervention to post-intervention as measured by ISS. | Baseline to end of active learning phase [week 4 for personalized intervention and week 6 for the general intervention]
  Bipolar symptoms will be measured using the Internal State Scale (ISS). The ISS is a 15 item self-report instrument using a visual analog line scale format (i.e. participant chooses from 0-100 on the scale to respond to each item). The scale contains four subscales (Activation, Well Being, Depression Index, and Perceived Conflict). Scores range from 0 to 1500 where higher scores represent higher severity of symptoms for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bress, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No